CLINICAL TRIAL: NCT04141423
Title: An Open Label, Multiple Ascending Dose Trial in Patients With T1DM to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Insulin Tregopil and to Evaluate the Postprandial Glucose Control With Different Meal Types in Comparison With Insulin Aspart
Brief Title: Evaluation of Pharmacokinetics , Safety, Tolerability and Pharmacodynamics of Biocon Insulin Tregopil
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part 1 completed. Part 2 not initiated
Sponsor: Biocon Limited (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TREGO-DM1-01-G-02
Record Dates: First submitted 2019-10-16; First posted 2019-10-28 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Type 1 Diabetes Mellitus (T1DM)
Keywords: Oral Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Indium-105

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tregopil 30 mg (Active Comparator): Dose level cohort with a sentinel dosing design
  Interventions: Drug: Tregopil
- Tregopil 45 mg (Active Comparator): Dose level cohort with a sentinel dosing design
  Interventions: Drug: Tregopil
- Tregopil 60 mg (Active Comparator): Dose level cohort with a sentinel dosing design
  Interventions: Drug: Tregopil
- Derived Dose level (Active Comparator): Derived Dose level cohort with a sentinel dosing design (60 mg fixed preprandial dose plus an additional 30 mg postprandial rescue dose, if required)
  Interventions: Drug: Tregopil

INTERVENTIONS:
Drug: Tregopil — Insulin Tregopil is recombinant human insulin modified by a single amphiphilic oligomer covalently linked via an amide bond to lysine at position 29 of the B-chain. This alters the physicochemical characteristics of the molecule, leading to enhanced stability and resistance to intestinal degradation following oral administration.
  Other Names: IN-105

SUMMARY:
Multi-centre, open label, multiple ascending dose trial in patients with type 1 diabetes mellitus

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multiple dose trial with two parts in patients with type 1 diabetes mellitus (T1DM). Part 1 consists of four cohorts with multiple ascending doses of insulin Tregopil and comprises a sentinel dosing design. Part 2 consists of a randomised, 2-treatment, crossover design with mixed meal tests (MMTs) of different compositions followed by parallel design titrated treatment period. Both parts include dosing during an in-house period and during a subsequent outpatient period.

ELIGIBILITY:
Inclusion Criteria (key criteria):

1. Male or female patient with diabetes mellitus type 1 on insulin therapy for at least 1 year before screening
2. Age between 18 and 64 years, both inclusive.
3. Body Mass Index (BMI) between 18.5 and 29.0 kg/m2, both inclusive.
4. Body weight between 60 kg and 100 kg, both inclusive and a stable weight +/- 5% for at least 3 months prior to screening (evaluated by patient history or medical history documents).
5. Beta-N-1-deoxy fructosyl haemoglobin (HbA1c) between 6.5 to 9%, both inclusive.
6. Total insulin dose of < 1.2 (I)U/kg/day.
7. Daily dose of prandial insulin analogues or regular human insulin not exceeding 70% of total daily insulin dose at screening.
8. Fasting C-peptide <= 0.20 nmol/L.
9. Daily dose of prandial insulin analogues or regular human insulin of at least 21 (I)U per day at screening.
10. Stable basal-bolus insulin regimen for at least 3 months prior to screening (stable as per Investigator's discretion).
11. Patients with experience in insulin titration and self-treatment of hypoglycemic events.
12. Considered generally healthy (apart from conditions associated with T1DM) upon completion of medical history and screening safety assessments including safety lab results, as judged by the Investigator.

Exclusion Criteria(key criteria):

1. Use of continuous subcutaneous insulin infusion (CSII) in the last 3 months prior to screening.
2. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
3. History of autoimmune disorders other than T1DM as judged clinically relevant by the Investigator (obtained by patient history), except a stable thyroid disorder treated with a stable dose of thyroxin.
4. Hospitalization for diabetic ketoacidosis during the previous 6 months.
5. More than one episode of severe hypoglycemia (as per American Diabetes Association classification) with seizure, coma or requiring assistance of another person during the past 6 months.
6. Hypoglycemic unawareness (defined as individuals with a score of 3 or more [reduced awareness and intermediate awareness] as assessed by the Clarke score).
7. Presence of clinically significant acute gastrointestinal (GI) symptoms (e.g. nausea, vomiting, heartburn or diarrhea) within 2 weeks prior to dosing, as judged by the investigator.
8. Presence of chronic GI disorders or conditions known to significantly alter the absorption of orally administered drugs or significantly alter upper GI or pancreatic function, as judged by the Investigator.
9. Patient with previous gastrointestinal surgery, except patients that underwent uncomplicated surgical procedures such as appendectomy, hernia surgery, biopsies, as wells as colonic- and gastric endoscopy.
10. Treatment with glucagon-like peptide 1 (GLP-1) receptor agonists within the last 12 weeks prior to screening visit.
11. The use of any prescribed medication that would interfere with trial endpoints or the safe completion of the trial procedures like e.g. warfarin, indomethacin or systemic non-selective ß-blocker, as judged by the investigator.
12. Any clinically significant abnormality in ECG or safety laboratory tests (liver function, renal function, hematology, urinalysis or any other laboratory result judged as clinically relevant by the investigator) at screening.
13. Clinically significant cardiovascular and/or cerebrovascular disease within 12 months before Screening, as judged by the Investigator.
14. Active proliferative retinopathy as confirmed by ophthalmoscopy / retinal photography examination performed (by a qualified person as per local legislation) within 6 months prior to screening.
15. Renal impairment with estimated Glomerular Filtration Rate (eGFR) < 60 mL

    * min/1.73m2 as defined by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
16. History of severe form of neuropathy or clinically significant cardiac autonomic neuropathy (CAN).
17. Patients who needed systemic (oral, intravenous, intramuscular) glucocorticoid therapy within 4 weeks prior to the screening visit OR expected of requiring during the study period.
18. Patients who have undergone pancreatectomy or pancreas/islet cell transplant or had any significant pancreatic disease that affects safety of the patient.
19. Inability or unwillingness to refrain from smoking and use of nicotine substitute products one day before and during the study.
20. Patients refusing/not capable to consume three major meals per day on routine basis.
21. If female, pregnancy or breast-feeding.
22. Women of childbearing potential who are not using a highly effective contraceptive method.
23. Men with non-pregnant partner(s) of childbearing potential not willing to use male contraception (condom) in addition to a highly effective contraceptive method until one month after last dosing.
24. Men of childbearing potential not willing to refrain from sperm donation for the duration of the study and for one month following last dose of study drug.
25. Men with pregnant partner not willing to use male contraception (condom) until one month after last dosing, in order to avoid exposure of the embryo/foetus to seminal fluid.
26. Patients unwilling to avoid heavy machinery work, driving within specified post dose interval during the study treatment period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Between screening (up to Day -21) and End of study ( up to Day 6)
  Number of patients with Adverse Events (Part I)
Laboratory safety parameters | Between screening (up to Day -21) and End of study ( up to Day 6)
  Number of patients with clinically significant changes in Laboratory safety parameters (Part I)
Physical examination | Between screening (up to Day -21) and End of study ( up to Day 6)
  Number of patients with clinically significant changes in Physical examination (Part I)
Vital signs, clinically | Between screening (up to Day -21) and End of study ( up to Day 6)
  Number of patients with clinically significant changes in Vital signs (Part I)
Hypoglycaemic events | Between screening (up to Day -21) and End of study ( up to Day 6)
  Number of patients with Hypoglycaemia events (Part I)
Hyperglycaemia events | Between screening (up to Day -21) and End of study ( up to Day 6)
  Number of patients with Hyperglycaemia events (Part I)
Electrocardiograms | Between screening (up to Day -21) and End of Treatment ( up to Day 6)
  Number of patients with clinically significant changes in Electrocardiogram (ECG) (Part I)
Adverse events (AEs) | Day of screening to Day 20 (Diary) and During follow up Via (Telephone)
  Number of patients with Adverse Events (Part II)
Hypoglycaemic events | Day of screening to Day 20 (Diary) and During follow up Via (Telephone)
  Number of patients with Hypoglycaemia events (Part II)
Hyperglycaemia events | Day of Run-in to Day 20 (Diary) and During follow up Via (Telephone)
  Number of patients with Hyperglycaemia events (Part II)
Laboratory safety parameters | Day of screening and Day 20
  Number of patients with clinically significant changes in Laboratory safety parameters (Part II)
Physical examination | Day of screening, Dosing day 1 and Day 20
  Number of patients with clinically significant changes in Physical examination (Part II)
Vital signs | Day of screening, Day1-6 and Day 20)
  Number of patients with clinically significant changes in Vital signs (Part II)
Electrocardiograms | Day of screening and Day 20
  Number of patients with clinically significant changes in Electrocardiogram (ECG) (Part II)
Anti-insulin Tregopil antibodies | Day -1 and Day 20
  Change in antibody levels (Part II)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) endpoint-Area under the insulin concentration curve(AUCins). | 0 to 1 hour
  Area under the insulin concentration curve (Part I)
PK endpoint-Area under the insulin concentration curve(AUCins). | 0 to 2 hour
  Area under the insulin concentration curve (Part 1)
PK endpoint-Area under the insulin concentration curve(AUCins). | 0 to 3 hour
  Area under the insulin concentration curve (Part I)
PK endpoint-Area under the insulin concentration curve(AUCins). | 0 to 4 hour
  Area under the insulin concentration curve (Part I)
PK endpoint-Area under the insulin concentration curve(AUCins). | Time zero to the last measurable concentration (6 hours)
  Area under from time zero to the last measurable concentration sampling time (Part I)
PK endpoint-Area under the insulin concentration curve(AUCins). | Day 1, Day 2, Day 6
  AUC from time zero to infinity (Part I)
PK endpoint-time to maximum observed insulin concentration (tmax) | Day 1, Day 2, Day 6
  Time to maximum observed insulin concentration (Part I)
PK endpoint-terminal elimination half-life calculated | Day 1, Day 2, Day 6
  Terminal elimination half-life calculated as t½=ln2/ λz (Part I)
PK endpoint-Area under the insulin concentration curve in the intended dosing interval (AUCins) | Day 1, Day 2, Day 6
  Area under the insulin concentration curve in the intended dosing interval (Part I)
PK endpoint-Insulin concentration at the end of treatment (Ctrough) | Day 1, Day 2, Day 6
  Insulin concentration at the end of treatment (Part I)
PK endpoint-Insulin concentration in plasma, tlag (lag time) | Day 1, Day 2, Day 6
  Time to first appearance of insulin concentration in plasma after dosing (Part I)
pharmacodynamics (PD) Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals on Day 1, 2 and 6 mixed meal tests | 0-1 hour
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals | 0-2 hour
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals | 0-3 hour
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals | -10 min-6 hour
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals | 0-6 hour
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration curve in the indicated time intervals | 0-1 hour
  Area under the plasma glucose concentration curve in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration curve in the indicated time intervals | 0-2 hour
  Area under the plasma glucose concentration curve in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration curve in the indicated time intervals | 0-3 hour
  Area under the plasma glucose concentration curve in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration curve in the indicated time intervals | 0-4 hour
  Area under the plasma glucose concentration curve in the indicated time intervals (Part I)
PD Endpoints-Area under the plasma glucose concentration curve in the indicated time intervals | 0-6 hour
  Area under the plasma glucose concentration curve in the indicated time intervals (Part I)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals | 0-1 hour
  Minimum plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals | 0-2 hour
  Minimum plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals | 0-3 hour
  Minimum plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals | 0-4 hour
  Minimum plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals | 0-6 hour
  Minimum plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-maximal plasma glucose concentration in the indicated time intervals | 0-2 hour
  Maximal plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-maximal plasma glucose concentration in the indicated time intervals | 0-4 hour
  Maximal plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-maximal plasma glucose concentration in the indicated time intervals | 0-6 hour
  Maximal plasma glucose concentration in the indicated time intervals (Part I)
PD Endpoints-maximal plasma glucose observed sampling period | -10 min-6 hour
  maximal plasma glucose observed sampling period (Part I)
PD Endpoints- ΔGmin minimum postprandial plasma glucose increment, absolute and percent | 0-6 hour
  Minimum postprandial plasma glucose increment, absolute and percent (Part I)
PD Endpoints- time to onset of action; time to decrease in PG of 5 mg/dL from baseline | 0 hour
  Onset of action; time to decrease in PG of 5 mg/dL from baseline (Part I)
Duration of action; | 0- 6 hour
  time from onset of action to increase in PG ≥ 180 mg/dL post meal or time to increase to baseline PG if baseline > 180 mg/dL (Part I)
Continuous glucose monitoring (CGM) profile | 6 days
  daily glycaemic control assessed d by mean (SD) glucose levels, percentage of time in normal range [70-180 mg/dL], percentage of time in hyperglycaemia range [>180 mg/dL], percentage of time in hypoglycaemic range (<70 mg/dL), percentage of readings in the range of 70-180 mg/dL (3.9- 10.0 mmol/L) per unit of time (Part I)
PK Endpoints- Maximum concentration recorded ( Day 1, 2,3,4,5,6,20) | 0-4 hours
  Maximum concentration recorded (Cmax) (Part II)
PK Endpoints-Area under the insulin concentration curve ( Day 1, 2,3,4,5,6,20) | 0-1 hours
  Area under the insulin concentration curve (AUC) (Part II)
PK Endpoints-Area under the insulin concentration curve ( Day 1, 2,3,4,5,6,20) | 0-2 hours
  Area under the insulin concentration curve (AUC) (Part II)
PK Endpoints-Area under the insulin concentration curve ( Day 1, 2,3,4,5,6,20) | 0-4 hours
  Area under the insulin concentration curve (AUC) (Part II)
PK Endpoints-Area under the insulin concentration curve ( Day 1, 2,3,4,5,6,20) | 0-6 hours
  Area under the insulin concentration curve (aspart) (AUC) (Part II)
PK Endpoints-Area under the insulin concentration curve ( Day 1, 2,3,4,5,6,20) | 0-last
  Area under the insulin concentration curve (AUC) (Part II)
PK Endpoints-Area under the insulin concentration curve ( Day 1, 2,3,4,5,6,20) | 0-∞
  Area under the insulin concentration curve (AUC) (Part II)
PK Endpoints- terminal elimination half-life calculated ( Day 1, 2,3,4,5,6,20) | Day 1, Day 2,Day 3,Day 4, Day5, Day 6, Day 20
  Terminal elimination half-life calculated as t½=ln2/ λz (Part II)
PK endpoint-time to maximum observed insulin concentration (tmax) ( Day 1, 2,3,4,5,6,20) | Day 1, Day 2,Day 3,Day 4, Day5, Day 6, Day 20
  Time to maximum observed insulin concentration (Part II)
PK Endpoints-Area under the insulin concentration curve ( Day 1, 2,3,4,5,6, 20) | Day 1, Day 2,Day 3,Day 4, Day5, Day 6, Day 20
  Area under the insulin concentration curve (AUC) (Part II)
PK endpoint-Insulin concentration at the end of treatment ( Day 1, 2,3,4,5,6, 20) | Day 1, Day 2,Day 3,Day 4, Day5, Day 6, Day 20
  Insulin concentration at the end of treatment (Ctrough) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-1 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GExc) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-2 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GExc) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-3 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GExc) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-4 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GExc) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6,20) | 0-6 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GExc) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-1 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GAUC) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-3 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GAUC) (Part II)
PD Endpoints-Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-4 hours
  Area under the plasma glucose concentration excursion from baseline (pre-meal) in the indicated time intervals (GAUC) (Part II)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-1 hours
  Minimum plasma glucose concentration in the indicated time intervals (Gmin) (Part II)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals ( Day 1, 2,3,4,5,6,20) | 0-3 hours
  Minimum plasma glucose concentration in the indicated time intervals (Gmin) (Part II)
PD Endpoints-minimum plasma glucose concentration in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-4 hours
  Minimum plasma glucose concentration in the indicated time intervals (Gmin) (Part II)
PD Endpoints-maximal plasma glucose concentration in the indicated time intervals ( Day 1, 2,3,4,5,6, 20) | 0-4 hours
  Maximal plasma glucose concentration in the indicated time intervals (Gmax) (Part II)
PD Endpoints -minimal PG concentration in observed sampling period ( Day 1, 2,3,4,5,6, 20) | 0 - 6 hours
  minimal PG concentration in observed sampling period (Part II)
PD Endpoints - maximal PG concentration in observed sampling period ( Day 1, 2,3,4,5,6, 20) | 0 - 6 hours
  maximal PG concentration in observed sampling period (Part II)
PD Endpoints - CGM profile | Day 1 to 20
  CGM profile

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH Hellersbergstraße 9 (Acting as Coordinating Investigator); Leona Plum Mörschel, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH Hellersbergstraße 9
Locations (1):
- Profil Mainz GmbH & Co. KG Malakoff-Passage,Rheinstraße 4C D-55116, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latres E, Plum-Moerschel L, Murugesan SMN, Lou O, Panda J, Marwah A, Samsonraj R, Gopu CL, Loganathan S, Athalye SN. An open-label, multiple ascending dose trial of orally administered insulin Tregopil in patients with type 1 diabetes mellitus to evaluate its pharmacokinetics, pharmacodynamics, safety and tolerability. Diabetes Obes Metab. 2025 Jun;27(6):3154-3164. doi: 10.1111/dom.16327. Epub 2025 Apr 10. PMID 40211481